CLINICAL TRIAL: NCT01306422
Title: A Two Stage, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Kinetics and Efficacy of Twice-Daily Repeat Intake of 1110 mg of Hoodia Gordonii Purified Extract (PYM50717)
Brief Title: Safety, Tolerability, Kinetics and Efficacy Study of Hoodia Gordonii Purified Extract (PYM50717)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Phytopharm (Industry); Covance (Industry)
Responsible Party: Leo Abrahamse, PhD, Unilever R&D Vlaardingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07044V
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Appetite Depressant; Overweight; Body Weight
Keywords: hoodia gordonii; energy intake; food intake; efficacy; body weight; functional food; plant extract; safety; steroid glycosides; tolerability
MeSH Terms: conditions — Anorexia; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Stage 2: Placebo (Placebo Comparator): Placebo product, twice-daily, 65 minutes before breakfast and dinner
  Interventions: Other: Placebo yogurt drink
- Stage 2: H.g.PE 1110 mg b.d. (Active Comparator): Hoodia gordonii Purified Extract (H.g.PE) formulated product (1110 mg), twice-daily, 65 minutes before breakfast and dinner
  Interventions: Other: Hoodia gordonii purified extract (H.g.PE)
- Stage 1: placebo, breakfast & dinner (Placebo Comparator): Placebo product, twice-daily for two days, 65 minutes before breakfast and dinner
  Interventions: Other: Placebo yogurt drink
- Stage 1: H.g.PE 1110 mg breakfast/dinner (Active Comparator): Hoodia gordonii purified extract (H.g.PE) formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and dinner
  Interventions: Other: Hoodia gordonii purified extract (H.g.PE)
- stage 1: Placebo breakfast/lunch (Placebo Comparator): Placebo product, twice-daily for two days, 65 minutes before breakfast and lunch
  Interventions: Other: Placebo yogurt drink
- Stage 1: H.g.PE 1110 mg breakfast/lunch (Active Comparator): Hoodia gordonii purified extract (H.g.PE) formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and lunch
  Interventions: Other: Hoodia gordonii purified extract (H.g.PE)

INTERVENTIONS:
Other: Hoodia gordonii purified extract (H.g.PE) — H.g.PE(1110 mg) formulated yogurt drink, twice-daily, 65 minutes before breakfast and dinner, for 15 days
  Other Names: PYM50717; H.g.PE; Hoodia gordonii Purified Extract
  Arms: Stage 2: H.g.PE 1110 mg b.d.
Other: Placebo yogurt drink — Placebo product (yogurt drink matching the H.g.PE extract formulated yogurt drink in nutritional composition and taste. Placebo is consumed twice-daily, 65 minutes before breakfast and dinner for 15 days.
  Arms: Stage 2: Placebo
Other: Placebo yogurt drink — Placebo product, twice-daily for two days, 65 minutes before breakfast and lunch
  Arms: stage 1: Placebo breakfast/lunch
Other: Placebo yogurt drink — Placebo product, twice-daily for two days, 65 minutes before breakfast and dinner
  Arms: Stage 1: placebo, breakfast & dinner
Other: Hoodia gordonii purified extract (H.g.PE) — H.g.PE formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and lunch
  Other Names: PYM50717; H.g.PE; Hoodia gordonii Purified Extract
  Arms: Stage 1: H.g.PE 1110 mg breakfast/lunch
Other: Hoodia gordonii purified extract (H.g.PE) — H.g.PE formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and dinner
  Other Names: PYM50717; H.g.PE; Hoodia gordonii Purified Extract
  Arms: Stage 1: H.g.PE 1110 mg breakfast/dinner

SUMMARY:
The objective of this clinical study was to assess the safety, tolerability, efficacy (effects on appetite scores, food intake) and plasma kinetics of Hoodia gordonii purified extract (H.g.PE), when consumed twice-daily for 2 or 15-days.

DETAILED DESCRIPTION:
A two stage randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, kinetics and efficacy of twice-daily repeat intake of formulated Hoodia gordonii purified extract (H.g.PE) (PYM50717) administered twice daily for 2 or 15 days to healthy, overweight females aged 18 to 50 years with a body fat of 25-45%.

Stage 1 (pilot): Placebo controlled, double blind comparison to assess the effect of timing of product administration (i.e. breakfast and lunch vs breakfast and dinner).

Stage 2 (main study): Placebo controlled double blind comparison with product administered with breakfast and dinner.

A total of 64 subjects were included in this study; stage 1: n=15, stage 2: n=49. Treatment groups in stage 2 were matched for percentage body fat.

Stage 1:

* H.g.PE formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and lunch (n = 4).
* Placebo product, twice-daily for two days, 65 minutes before breakfast and lunch (n = 3).
* H.g.PE formulated product (1110 mg), twice-daily for two days, 65 minutes before breakfast and dinner (n = 5).
* Placebo product, twice-daily for two days, 65 minutes before breakfast and dinner (n = 3).

Stage 2:

* H.g.PE formulated product (1110 mg), twice daily (n=25)for 15 days
* Placebo product , twice daily (n=24),for 15 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between the ages of 18 and 50 years.
* Body fat between 25% and 45% as assessed by Dual Energy X-ray absorptiometry (DEXA) scan at Screening.
* Stable body weight for at least two months prior to Screening (weight loss or gain >5% was considered unstable).
* Regularly consumed at least three meals per day, including breakfast.
* Agreed to abstain from strenuous exercise throughout the entire study.

Exclusion Criteria:

* Subjects who were pregnant, lactating or were not willing to use two contraceptives (including at least one barrier contraceptive) starting at least 14 days before study product administration (Day 1) and until at least 30 days following study product administration (except subjects who were surgically sterilized or were more than one year post-menopausal).
* Subjects who were taking any prescription or over the counter medications (with the exception of hormonal contraceptives) (including supplements, especially as related to weight management [eg, ephedrine, caffeine, synephrine]) within one week prior to Visit 2 (Day 1), or antibiotics <3 months prior to Day 1, or planned to do so during the course of the study.
* Smokers, or ex-smokers who smoked any cigarettes in the past six months prior to study product administration and/or who used another form of nicotine-containing product.
* Fasting blood glucose > 7 mmol/L (126 mg/dL) at Screening.
* Psychiatric disorders that could have interfered with the subject's compliance to the requirements of the protocol, at the discretion of the Investigator.
* Used or planned to use any medically prescribed diet or weight-loss diet or made any attempt to control diet at Screening and during the entire study.
* Strenuous exercise >5 hours per week (eg, sports).
* Restrained eating behavior determined by a score of ≥16 on the Revised Restraint Scale
* a low score on the Food Action Rating Scale

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 2 and 15 day repeat consumption of Hoodia gordonii Purified Extract (H.g.PE) | 41 days
  Safety and tolerability (Adverse Events (AEs), vitals signs, Electrocardiogram (ECG), laboratory assessments) of twice daily consumption of 1110 mg of formulated Hoodia gordonii purified extract (H.g.PE) consumed over a period of 2 or 15 days were assessed up to 41 days after start of the intervention
Efficacy of 15-day repeat consumption of H.g.PE | 15 days
  Efficacy of twice daily consumption of 1110 mg of formulated H.g.PE during 15-day repeat intake was assessed. Appetite scores, ad libitum energy intake, body weight and body composition were assessed during the 15-day intervention.

SECONDARY OUTCOMES:
Assessment of the pharmacokinetics of PYM50057 a marker of the steroid glycosides in H.g.PE | 41 days
  Kinetic parameters were calculated on Days 5 and 19 based on the individual plasma concentration-time profiles of the steroid glycoside, PYM50057. Maximum measured plasma concentration (Cmax), time of Cmax (tmax), area under the concentration-time curve (AUC), apparent terminal phase rate constant (Kel), absorption rate constant (Ka),the apparent first order elimination rate constant (λz) and the overall apparent elimination half-life (t1/2) were assessed. Samples were taken up to 41 days after start of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Mandarino, MD, Principal Investigator — Covance CRU, Madison WI; Leo Abrahamse, PhD, Study Chair — Unilever R&D Vlaardingen
Locations (1):
- Covance CRU, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Blom WA, Abrahamse SL, Bradford R, Duchateau GS, Theis W, Orsi A, Ward CL, Mela DJ. Effects of 15-d repeated consumption of Hoodia gordonii purified extract on safety, ad libitum energy intake, and body weight in healthy, overweight women: a randomized controlled trial. Am J Clin Nutr. 2011 Nov;94(5):1171-81. doi: 10.3945/ajcn.111.020321. Epub 2011 Oct 12. PMID 21993434